CLINICAL TRIAL: NCT02840734
Title: Kinesio Taping and Muscular Function in Obese Adults
Brief Title: Effects of Kinesio Taping on Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Suk H. Lee, Program Director & Associate Professor, Texas A&M University San Antonio
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Tamusa
Record Dates: First submitted 2016-05-06; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Kinesio taping; Obese adults; Muscular function; Fatigue
MeSH Terms: conditions — Obesity; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio taping (Experimental): All subjects wore an eye mask and the taped leg was covered by clothes for preventing subjects and researchers from identifying different tapings due to double-blinding. Subjects layed down on the mat in a supine position with the hip flexed 30º and the knee flexed 60º. Y type tape was applied from a point 10 cm below the anterior superior iliac spine, bisected at the junction between quadriceps femoris tendon and the patella, ending at its inferior side. And another Y type tape was applied from the tibial tuberosity, bisected at the junction between patella tendon and the patella, ending at its superior side. The first 5 cm tape was not stretched and acted as the anchor. I type tapes were applied downward and inward to the superior and inferior meniscus of the patella respectively.
  Interventions: Other: Kinesio taping
- Placebo taping (Placebo Comparator): Placebo tapes (3M tape) were applied with same method with Kinesio taping.
  Interventions: Other: Kinesio taping
- No taping (No Intervention): In case of the no taping condition, the subject was treated along the same procedure which was closed subject's eyes with eye mask and covered the legs with clothes although applied anything on their legs. It might be able to minimize the error, because the researchers did not realize which condition the subject had.

INTERVENTIONS:
Other: Kinesio taping — This study was conducted in a randomized crossover double-blind design. Each subject was tested for muscular power, strength, endurance, and fatigue of the lower extremities under three conditions: 1) NT (no taping), 2) PT (placebo taping, 3M tape) and 3) KT (Kinesio taping). For allocation of treatment sequence, the participants drew straws for which treatment first (each treatment indicated different numbers).
  Other Names: Placebo taping
  Arms: Kinesio taping; Placebo taping

SUMMARY:
This study investigated the immediate effects of Kinesio taping on muscular power, strength, endurance, and lower limb fatigue when taping is applied to rectus femoris and around the patella of obese adults based on Kinesio taping techniques.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover, and clinical trial. Ethical approval was obtained from the University's Institutional Review Board (#2015-51). Participants were recruited by flyers posted on the University campus. Informed consent was completed by all participants prior to the study procedures. The subjects were obese college students. A total of 13 subjects, four males and nine females (mean age of 24.38 ± 3.01 years, mean percent body fat of 39.10 ± 6.91 % [male: 41.93 ± 7.47 %, female: 38.16 ± 6.91 %]), were enrolled this study. All subjects underwent three different trials which include no taping (NT), placebo taping (PT), and Kinesio taping (KT). All individuals were assessed for peak and mean power, muscular strength, endurance, and muscle fatigue after each condition.

ELIGIBILITY:
Inclusion Criteria:

* percent body fat of 25 % in males, 30 % in females or more

Exclusion Criteria:

* lower limb surgery within previous 6 months
* presence of any other lower limb joint diseases such as degenerative arthritis, rheumatoid arthritis.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Physique characteristic | 1 week (Each subject was measured their anthropometrics variables in an Initial visit the LAB for trial)
  - variables:(1) Body weight and height (Detecto DR400C platform scale (Webb City, MO) and Seca S-214 height rod (Hanover, MD), respectively), (2) Waist and hip circumference (Gulik tape measure), (3) % Body fat (bioelectrical impedance analysis, RJL Quantum X).

SECONDARY OUTCOMES:
muscular power | 4 weeks (30 minutes after applied each trial)
  Peak power and mean power were measured with automatic Power cycle (Powercycle, USA). The subjects started from rest and accelerated maximally for approximately 3-4 seconds. Data was recorded for 6.5 pedal revolutions, and the increase in kinetic energy resulting from the acceleration of the ergometer flywheel was averaged over every pedal revolution and used to calculate power. The highest power and mean power (average two of the highest values) recorded during a pedal revolution was defined as Pmax and Pmean respectively.
muscular strength | 4 weeks (30 minutes after applied each trial)
  Assessment of muscle strength was measured by Muscle Testing system. A hand-held dynamometer (Lafayette, USA) used to measure isometric knee extensor and flexor strength. Specifically, subjects were seated on a table in supine position, with the knee and hip positioned at 90º. The subjects were instructed to remain seated and place both hands on the table. The dynamometer force pad placed just proximal to the ankle joint, the knee extensor strength was quantified in pound force. All subjects performed two maximal trials for 3 to 5 seconds with a 30 seconds rest interval. The higher value of two trials was recorded.
muscle fatigue | 4 weeks (immediately after be completed each trial)
  To measure the sensation of lower limb muscle fatigue, subjects' subjective feelings were evaluated using a Visual Analogue Scale (VAS). A 100 mm VAS (on a 0-10 scale) was used, ranging from "not in the least (0)" on the left to "extremely (10)" on the right end. Participants were asked to score the amount of lower limb muscle fatigue experienced before and immediately after each trial.

CONTACTS AND LOCATIONS:
Overall Officials: Sukho Lee, Ph.D., Principal Investigator — Texas A&M University San Antonio

IPD SHARING:
Plan to Share IPD: Undecided